CLINICAL TRIAL: NCT01052675
Title: Pharmacological, Clinical and Statistical Assessment of a New Tool Available for Pharmacodependence Report Evaluation
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/07/10-C
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Drug Abuse; Drug Dependence
Keywords: Drug and substance problematic use, abuse or dependence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacodependance cases: Case report from one of the French CEIP for drug and substance problematic use, abuse or dependence except alcohol and tobacco.

SUMMARY:
In France, the Afssaps is the body in charge of the evaluation of pharmacodependance. In order to fulfil its mission, the Afssaps has created a network of 11 Centres for Evaluation and Information on Pharmacodependance (CEIP), coordinated by the Drugs and Psychotropics Unit. Pharmacodependence notifications issued by professionals are collected by each Centre which evaluates them. Nantes' CEIP created an original tool to harmonize case reporting and make it possible to homogeneously evaluate the seriousness of pharmacodependence cases as each CEIP had his own way of analysing his cases. The aim of this study is to assess this tool.

ELIGIBILITY:
Inclusion Criteria:

* case report from one of the French CEIP for drug and substance problematic use, abuse or dependence except alcohol and tobacco.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pharmacodependent patients
Sampling Method: Probability Sample
Enrollment: 3180 (Actual)
Dates: Start 2008-01-03 (Actual); Primary Completion 2011-06-14 (Actual); Study Completion 2013-09-15 (Actual)

PRIMARY OUTCOMES:
Psychometrics properties Evaluation of the new questionnaire centered on addiction to medicine . | At the beginning of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jolliet Pascale, MD, Study Director — Nantes's University Hospital
Locations (10):
- France (10):
  - Hôpital Pellegrin, Bordeaux
  - CHRU de Caen, Caen
  - CHU de Grenoble, Grenoble
  - Centre Antipoison - Centre de Pharmacovigilance, Lyon
  - Hôpital Salvator, Marseille
  - Hôpital Lapeyronie, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Fernand Widal, Paris
  - Faculté de médecine, Toulouse

REFERENCES:
- [Derived] Victorri-Vigneau C, Hardouin JB, Rousselet M, Gerardin M, Guerlais M, Guillou M, Bronnec M, Sebille V, Jolliet P; French Addictovigilance Network. Multicentre study for validation of the French addictovigilance network reports assessment tool. Br J Clin Pharmacol. 2016 Oct;82(4):1030-9. doi: 10.1111/bcp.13044. Epub 2016 Jul 28. PMID 27302554